CLINICAL TRIAL: NCT02843841
Title: Polyclonal Antilymphocyte Globulin (ATG) & Intestinal Immune Barrier After Kidney Transplantation
Acronym: GABII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2014/221
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-07

CONDITIONS: Disorder Related to Renal Transplantation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATG group (Other): Renal transplant Patients from Nephrology department of the University Hospital of Besancon receiving induction immunosuppressive therapy of polyclonal antilymphocyte globulin (ATG-Fresenius®) as recommended.
  Intervention = blood and fecal sample
  Interventions: Other: Blood and fecal sample.
- Anti-CD25 group (Other): PRenal transplant Patients from Nephrology department of the University Hospital of Besancon receiving induction immunosuppressive therapy of anti-CD25 monoclonal antibodies (basiliximab SIMULECT®) as recommended.
  Intervention = blood and fecal sample
  Interventions: Other: Blood and fecal sample.

INTERVENTIONS:
Other: Blood and fecal sample. — Blood (28 ml) and fecal sample at day 0, 4 days, 3 months and one year after transplantation

SUMMARY:
The prevention of allograft rejection in kidney transplantation requires administering to the patient an immunosuppressive regimen of induction. The induction strategy is based on an injection of polyclonal anti-lymphocyte globulin (ATG-FLAG or fresenius®) driving a lymphocyte lysis, or an injection of monoclonal antibodies directed against non-lymphopenic the α chain of the IL-receptor 2 (anti-CD25 antibody, basiliximab), by immunological risk patients. Our group showed a significant increase in death rates in transplant patients with lymphopenia CD4 continued beyond 2 years of transplantation. This excess mortality is related to complications following chronic inflammation observed in some patients lymphopenic.

Preliminary studies have shown that the induced lymphodéplétion ATG appears to be accompanied by an increase of the bacterial products in the blood of transplanted since a significant increase in the sCD14 is observed in these patients one year. We also observed increased concentrations of LPS in patients in the ATG group. This could indicate a secondary bacterial intestinal translocation to a weakening of intestinal immunity linked to the ATG.

The main objective of the study is to assess the impact of anti-lymphocyte globulin polyclonal on intestinal permeability, estimated by the rate lipopolysaccharide (LPS, a constituent of the cell wall of Gram-negative bacteria) blood after kidney transplantation.

The secondary objectives are to evaluate bacterial translocation, the effect of bacterial translocation on structural and metabolic functions of the intestinal epithelium, chronic inflammation, immune reconstitution, regeneration, activation and proliferation of T lymphocytes, the polymorphism of the LPS receptor that causes the activation of innate immunity and the composition of the intestinal microbiota.

The study population consists of renal transplant patients of Nephrology of the University Hospital of Besancon. Patients will be divided into 2 groups according to induction immunosuppressive therapy prescribed the day of renal transplantation as part of their usual care, ie treatment with anti-lymphocyte globulin polyclonal (ATG-Fresenius®) or antibody treatment monoclonal anti-CD25 (basiliximab Simulect). The patient group treated with anti-CD25 antibody will serve as a control group (no depletion of the immune system) to the group of patients treated with ATG.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years included
* Postmenopausal women for at least 24 months, sterilized surgically, or for women of childbearing age, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, method of double-barrier contraceptive patches)
* Participation in the study ORLY East
* Signature of informed consent for participation indicating that the subject has understood the purpose and procedures required by the study and agrees to participate in the study and comply with the requirements and limitations inherent in this study
* Join a French social security or receiving such a plan

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Topic unlikely to cooperate in the study and / or low early cooperation by the investigator
* Without health insurance Topic
* Pregnant woman
* Inability to understand the reasons for the study; psychiatric disorders judged by the investigator to be incompatible with the inclusion in the study
* Infectious episode with need for hospitalization older than 1 month
* Active infection by the virus of hepatitis B and / or C
* Active infection by HIV or not
* Patients with inflammatory bowel disease (IBD)
* Patients who have undergone total colectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03-01 (Actual); Study Completion 2017-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum LPS rate | 1 year
  LPS serum levels of kidney transplant patients treated with ATG evaluated by liquid chromatography coupled with mass spectroscopy before transplantation and 1 year after transplantation compared to renal transplant patients treated with anti-CD25 antibody.

SECONDARY OUTCOMES:
The serum levels of LPS. | 0, 4 days and 3 months after transplantation
  The results will be correlated to clinical data reported during the first year following the day of transplantation, namely: CMV disease, severe opportunistic infections bacterial infections, atherosclerotic events, dialysis back, patient treatment (antibiotics, standard treatment at the time of sampling).
The serum levels of translocation marker and intestinal integrity (CD14, citrulline, LBP, CETP, PLTP, IFABP) | 0, 4 days, 3 months and one year after transplantation
  All secondary endpoints will be measured at 0, 4 days, 3 and 12 months after transplantation. The results will be correlated to clinical data reported during the first year following the day of transplantation, namely: CMV disease, severe opportunistic infections bacterial infections, atherosclerotic events, dialysis back, patient treatment (antibiotics, standard treatment at the time of sampling).
The serum levels of inflammatory cytokines (IL-1β, IL-6, TNF-α, IL-8, IL 12, CRP) | 0, 4 days, 3 months and one year after transplantation
  All secondary endpoints will be measured at 0, 4 days, 3 and 12 months after transplantation. The results will be correlated to clinical data reported during the first year following the day of transplantation, namely: CMV disease, severe opportunistic infections bacterial infections, atherosclerotic events, dialysis back, patient treatment (antibiotics, standard treatment at the time of sampling).
The serum levels of regeneration cytokines (IL-7, IL-15 and IL-22) | 0, 4 days, 3 months and one year after transplantation
  All secondary endpoints will be measured at 0, 4 days, 3 and 12 months after transplantation. The results will be correlated to clinical data reported during the first year following the day of transplantation, namely: CMV disease, severe opportunistic infections bacterial infections, atherosclerotic events, dialysis back, patient treatment (antibiotics, standard treatment at the time of sampling).
Serum percentage of CD8+CD57+CD28- LT, CD31+CD4+CD45RA+ LT, Lin-CD34+CD45+CD10+CD38+CD117-CD45RA+ LT, CD3+CD4/8+HLADR+CD38+ LT, Ki67 | 0, 4 days, 3 months and one year after transplantation
  All secondary endpoints will be measured at 0, 4 days, 3 and 12 months after transplantation. The results will be correlated to clinical data reported during the first year following the day of transplantation, namely: CMV disease, severe opportunistic infections bacterial infections, atherosclerotic events, dialysis back, patient treatment (antibiotics, standard treatment at the time of sampling).
TLR-4 polymorphism | 0, 4 days, 3 months and one year after transplantation
  All secondary endpoints will be measured at 0, 4 days, 3 and 12 months after transplantation. The results will be correlated to clinical data reported during the first year following the day of transplantation,
The composition of the intestinal microbiota. | 0, 4 days, 3 months and one year after transplantation
  All secondary endpoints will be measured at 0, 4 days, 3 and 12 months after transplantation. The results will be correlated to clinical data reported during the first year following the day of transplantation,

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Bamoulid, Dr., Principal Investigator — Besancon University Hospital - Nephrology departement
Locations (1):
- Besancon University Hospital, Besançon, France, France

IPD SHARING:
Plan to Share IPD: No